CLINICAL TRIAL: NCT03269149
Title: Effects of Adapted Tango on African-American Women Caregivers of Alzheimer's Disease Patients
Brief Title: Tango for Alzheimer's Disease Patients' Caregivers
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Principal Investigator, Madeleine Eve Hackney, Asstant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00097348
Record Dates: First submitted 2017-08-30; First posted 2017-08-31 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Alzheimer's Disease
Keywords: Alzheimer's disease; African-American Women; Caregivers; Tango; Dance-based intervention
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adapted Tango Dance (Experimental): 20 improvisational, 90-minute adapted tango dance sessions over a 12-week period.
  Interventions: Other: Adapted Tango Dance
- Educational Control (Active Comparator): Participants will take part in at least 20 educational lectures offered twice per week over 12 weeks.
  Interventions: Behavioral: Educational lectures

INTERVENTIONS:
Other: Adapted Tango Dance — 20 improvisational, 90-minute adapted tango dance sessions over a 12-week period. Classes begin with a 20-minute standing warm-up followed by partnering and rhythmic exercises. Next, novel step elements are introduced and participants will be taught how to combine the new steps with previously learned steps via improvisation. Caregivers will dance with each other or undergraduate /graduate student volunteers. Music will be played throughout classes and artistic expression, i.e., attention to aesthetics, and improvisation, will be encouraged.
  Arms: Adapted Tango Dance
Behavioral: Educational lectures — Participants will take part in at least 20 educational lectures offered twice per week over 12 weeks. Classes will also be 1.5 hours long and will involve lecture, partnered and group learning and extensive Q&A will be encouraged.
  Arms: Educational Control

SUMMARY:
The goal of the project is to determine the extent to which indices of inflammatory biomarkers, cognition and mood, are influenced by a partnered, dance-based intervention vs control condition in African American (AA) female family caregivers, at high risk for Alzheimer's disease (AD).

DETAILED DESCRIPTION:
The importance of informal family caregiving in Alzheimer's disease (AD) is well-established. African-American caregivers are most often middle aged adult children of AD patients (vs. spouses), women, and are at higher risk for chronic health problems. AD lifestyle interventions offer an alternative to medication, and are generally affordable, accessible, and adaptable to the lives of caregivers. To date, most non-pharmaceutical interventions have focused on exercise and nutrition, both of which have proven to be highly successful in conferring AD related benefits and decreasing AD risk.

The goal of the project is to determine the extent to which indices of inflammatory biomarkers, cognition and mood, are influenced by a partnered, dance-based intervention vs control condition in African American (AA) female family caregivers, at high risk for Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

* Women family caregivers from the Emory ADRC and Dr. Wharton's studies of Alzheimer's disease (AD) caregivers
* Parental diagnosis 'probable AD'
* African-American
* 45-65 years of age

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Females
Enrollment: 60 (Estimated)
Dates: Start 2017-09-19 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in interleukin-7 | Before and after the intervention / control at least 20 times during 12 weeks
  45 mL blood will be acquired before and after the intervention to measure the inflammatory and stress marker levels
Change in interleukin-8 | Before and after the intervention / control at least 20 times during 12 weeks
  45 mL blood will be acquired before and after the intervention to measure the inflammatory and stress marker levels
Change in interleukin-9 | Before and after the intervention / control at least 20 times during 12 weeks
  45 mL blood will be acquired before and after the intervention to measure the inflammatory and stress marker levels
Change in Interleukin-10 | Before and after the intervention / control at least 20 times during 12 weeks
  45 mL blood will be acquired before and after the intervention to measure the inflammatory and stress marker levels
Change in interferon induced protein 10 | Before and after the intervention / control at least 20 times during 12 weeks
  45 mL blood will be acquired before and after the intervention to measure the inflammatory and stress marker levels
Change in macrophage derived chemokine | Before and after the intervention / control at least 20 times during 12 weeks
  45 mL blood will be acquired before and after the intervention to measure the inflammatory and stress marker levels
Change in monocyte chemoattractant protein 1 | Before and after the intervention / control at least 20 times during 12 weeks
  45 mL blood will be acquired before and after the intervention to measure the inflammatory and stress marker levels
Change in transforming growth factor alpha | Before and after the intervention / control at least 20 times during 12 weeks
  45 mL blood will be acquired before and after the intervention to measure the inflammatory and stress marker levels
Change in tumor necrosis factor alpha | Before and after the intervention / control at least 20 times during 12 weeks
  45 mL blood will be acquired before and after the intervention to measure the inflammatory and stress marker levels
Change in C-reactive protein | Before and after the intervention / control at least 20 times during 12 weeks
  45 mL blood will be acquired before and after the intervention to measure the inflammatory and stress marker levels
Change in serum amyloid protein | Before and after the intervention / control at least 20 times during 12 weeks
  45 mL blood will be acquired before and after the intervention to measure the inflammatory and stress marker levels

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  The MoCA test is a 30-point test that assesses several cognitive domains. The short-term memory recall task (5 points) ; Visuospatial abilities are assessed using a clock-drawing task (3 points) and a three-dimensional cube copy (1 point); executive functions are assessed using an alternation task adapted from the trail-making B task (1 point), a phonemic fluency task (1 point), and a two-item verbal abstraction task (2 points). Attention, concentration and working memory are evaluated using a attention task (target detection using tapping; 1 point), a serial subtraction task (3 points), and digits forward and backward (1 point each). Language is assessed using a confrontation naming task with low-familiarity animals (3 points), repetition of two syntactically complex sentences (2 points), and the aforementioned fluency task. Finally, orientation to time and place is evaluated (6 points).
Change in the Tower of London test | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  The Tower of London test is used for the assessment of executive functioning specifically to detect deficits in planning. It is related to the classic problem-solving puzzle known as the Tower of Hanoi.The test consists of two boards with pegs and several beads with different colors. The examiner uses the beads and the boards to present the examinee with problem-solving tasks. The performance of the examinee is compared to representative samples of individuals of the same age to derive hypotheses about the person's executive cognitive ability.
Change in the Stroop interference test | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  The Stroop test is to name the color in which a word is printed, ignoring the word itself. The Stroop Test is used to assess the ability to inhibit cognitive interference that occurs when the processing of a specific stimulus feature impedes the imultaneous processing of a second stimulus attribute, well-known as the Stroop Effect. Total time needed for each card is the outcome variable.
Change in Trails B test | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  Trail Test is a neuropsychological test of visual attention and task switching. It consists of two parts in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The time taken to complete the test is used as the primary performance metric.The test is sensitive to detecting cognitive impairment.
Change in Digit Span test | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  The Digit Span test is either conducted verbally or using a computer program. A sequence of numbers is shown or read out to the participant. The participant is then told to repeat the numbers that were shown or read to them. This process continues until the participant can no longer remember either the full sequence of numbers or the correct order.The Digit Span test is scored by the amount of numbers the participant was able to remember in each test. The scorer must add the total number of correct sequences, backwards and forwards.
Change in Buschke Selective Reminding Test | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  The Buschke Selective Reminding Test (SRT) is a test designed to measure verbal learning and memory through the use of a list-learning procedure over multiple trials. The adult SRT involves reading the subject a list of 12 unrelated words and then having the subject immediately recall as many of these 12 words as possible. Every trial after the first involves selectively presenting only those words in which the subject did not recall on the immediately preceding trial. The selective reminding trials proceed in this manner until the subject is able to correctly recall all 12 words on three consecutive trials, or until 12 trials have been completed. Scoring of the test has been automated according the instructions of Buschke.
Change in Reverse Corsi Blocks test | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  The Corsi block-tapping test is a psychological test that assesses visuo-spatial short term working memory. It involves mimicking a researcher as he/she taps a sequence of up to nine identical spatially separated blocks. The sequence starts out simple, usually using two blocks, but becomes more complex until the subject's performance suffers. This number is known as the Corsi Span, and averages about 5 for normal human subjects.
Change in Brooks spatial memory test | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  Brooks spatial memory task (BSMT): In the BSMT, the participant visualizes a 4x4 matrix in which the location of numbers 1 through 8 is described. Participants practice with 3 instructions and progress up to 8 instructions. All levels are completed regardless of errors. Percentages correct (out of 50) will be used for analysis.
Change in the Body position spatial task (BPST) | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  Body position spatial task (BPST) measures whole body knowledge of spatial position and ability to navigate in a remembered path. The examiner verbally and visually demonstrates combinations of 5 possible moves: step forward, step left, step right, quarter turn left, and quarter turn right. The examiner begins with 2 moves and progresses up to 9 moves, with 2 trials per level. Participants continue to the next level if one trial is correctly performed. The test ends when participants miss both trials of a level. Span length and number of correct trials are variables.
Change in Fullerton Advanced Balance Scale | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  The Fullerton Test is mainly intended to identify highly-active older adults who are at an increased risk to experience fall-related injuries due to sensory impairments. The test uses both dynamic and static balance under different situations to identify balance deficits in older adults. The test includes the following: 10 performance based activities in both static and dynamic phases; Score of 0-40/40 points possible (higher scores are better); tems scored on a 5 point ordinal scale (0-4).
Change in 30-second chair stand | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  The 30 second chair test is administered using a folding chair without arms, with seat height of 17 inches (43.2 cm). The 30 second chair stand involves recording the number of stands a person can complete in 30 seconds.
Change in gait speed | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  Assesses walking speed in meters per second over a short duration . The individual is instructed to walk a set distance (6 meters, 10 meters, etc). Time is measured while the individual walks the set distance (often the individual is given space to accelerate to his/her preferred walking speed (this distance is not included when determining speed). The distance covered is divided by the time it took the individual to walk that distance.
Change in Positive Aspects of Caregiving (PAC) Scale | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  The 9-item PAC scale will be administered to the caregivers. Each item is scored on a 5-point Likert scale: disagree a lot (1), disagree a little (2), neither agree nor disagree (3), agree a little (4), and agree a lot (5). The overall PAC score, comprising all nine items, ranges from 9 to 45-a higher score reflects a more positive perception of the caregiving experience.
Change in Pearlin Caregiver Stress Scale | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  Pearlin Caregiver Stress Scale topics include primary stressors (cognitive status, problematic behavior, overload, relational deprivation), secondary role strains family conflict, job-caregiving conflict, economic strains), secondary instrapsychic strains (role captivity, loss of self, caregiving competence, personal gain) and mediators (management of situation, management of meaning, management of distress, expressive support). Fifteen 3-point to 5-point scales.
Change in the Zarit Burden Interview | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  The Zarit Burden Interview, a caregiver self-report measure is a 22-item self-report inventory that examines burden associated with functional/behavioral impairments and the home care situation. Each question is scored on a 5 point Likert scale ranging from 0 (Never) to 4 (Nearly Always).. Total scores range from 0 (low burden) to 88 (high burden).
Change in the Center for Epidemiologic Studies Depression Scale (CES-D) | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  The CESD-R is a screening test for depression and depressive disorder. The 20 items in CESDR scale measure symptoms of depression in nine different groups as defined by the American Psychiatric Association. The response values for each question are:
  Not at all or less than one day = 0 1-2 days = 1 3-4 days = 2 5-7 days = 3 Nearly every day for 2 weeks = 4 The Total CESD-R Score is calculated as a sum of responses to all 20 questions.
Change in DEMQOL: Dementia Quality of Life measure (Carer v4) | Before and after the intervention / control, offered twice per week, at least 20 times during 12 weeks
  DEMQOL is a 29-item scale, plus one global item ("Overall, how would you rate your quality of life?") that measures 5 domains of QOL: Positive Affect (6 items), Negative Affect (11 items), Feelings of Belonging (3 items), Self-esteem (4 items), and Sense of Aesthetics (5 items). The DQoL yields scores on 5 subscales but subscale scores are not summed to reach an overall or global measure of QOL.

CONTACTS AND LOCATIONS:
Overall Officials: Madeleine Hackney, Principal Investigator — School Of Medicine, Emory University
Locations (1):
- Atlanta VA Medical Center, Emory University, Executive Park, Wesley Woods, Atlanta, Georgia, United States

DOCUMENTS (1):
  • Informed Consent Form (2019-05-16): https://cdn.clinicaltrials.gov/large-docs/49/NCT03269149/ICF_000.pdf